CLINICAL TRIAL: NCT02389920
Title: Multicenter, PhaseⅣ, Open Label Trial of Nilotinib in Adult Patients Diagnosed Philadelphia Chromosome Positive(Ph+) Chronic Myeloid Leukemia in CP/AP Intolerant to Dasatinib
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Chul Won Jung, Samsung Medical Center, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-01-112
Record Dates: First submitted 2015-03-11; First posted 2015-03-17 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Leukemia, Chronic Myeloid
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — nilotinib

ARMS (1):
- Nilotinib (Experimental): nilotinib 400mg BID for 12 months
  Interventions: Drug: Nilotinib

INTERVENTIONS:
Drug: Nilotinib

SUMMARY:
Describe the purpose of the study: This study aims to evaluate the improvement of Dasatinib-related adverse events and to evaluate the treatment effect and safety by measuring the genetic response of nilotinib with nilotinib 400mg BID for 12 months in Philadelphia chromosome-positive chronic myeloid leukemia patients intolerant to Dasatinib.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women ≥ 19 years old
2. Performance status (ECOG) of 0, 1, or 2
3. Chronic phase or accelerated phase chronic myeloid leukemia being treated for more than two weeks, switch to nilotinib.
4. Appropriate target organ function defined as;

   - Bilirubin < 1.5 X ULN- Liver function test, AST (SGOT) and ALT (SGPT) < 2.5 X ULN- Creatinine < 1.5 X ULN- Serum amylase and lipase ≤ 1.5 X ULN- Alkaline phosphatase ≤ 2.5 X ULN (only if not related to tumor)
5. Women of childbearing potential must have a negative pregnancy test (urine or serum) within 7 days prior to the start of study drug administration.
6. Should have laboratory results as follows.

   - Potassium ≥ LLN- Magnesium ≥ LLN- Phosphorus ≥ LLN
7. Voluntary, signed and dated informed consent prior to any study procedures being performed

Exclusion Criteria:

1. Subjects with the T315I mutation
2. Mutation known to be associated with low sensitivity to nilotinib(e.g., Y253H, E255K, E255V, F359V),
3. Cardiac function abnormalities as follows are found.

   * FEVI < 45% or less than lower limit of normal of each center on ECG
   * QT interval cannot be measured on ECG
   * Complete right bundle branch block
   * Using a ventricular pacemaker
   * Congenital long QT syndrome or family history of long QT syndrome
   * Past or present clinically significant ventricular or atrial tachycardia
   * Clinically significant bradycardia at rest (< 50 beats/min)
   * Regardless of toxicity after Dasatinib intake, QTc > 480 msec (using the QTcF formula) at baseline ECG. If QTcF > 480 msec and electrolytes are not within the normal range, it is necessary to correct electrolytes and re-assess the patient's QTc. According to the result of QTc, the investigator makes a decision on the patient's enrollment.
   * Myocardial infarction within 12 months prior to the start of the study
   * Other clinically significant heart disease (e.g., unstable angina, congestive heart failure or uncontrolled hypertension)
4. Cytopathologically confirmed central nervous system lumbar puncture (spinal tapping is not needed if it is not suspected of association with central nervous system)
5. Severe or uncontrolled disease (e.g., uncontrolled diabetes mellitus, active or uncontrolled infection)
6. History of significant congenital or acquired, bleeding disorder unrelated to cancer
7. 25% or more of bone marrow has been treated with prior radiotherapy
8. Not recovered from prior surgery or having a major surgery within 4 weeks from Day -1 of the study
9. Treated with other investigational product within 30 days
10. History of noncompliance with medical treatment or unable to voluntarily provide the written signed and dated informed consent
11. Other primary cancer which is currently clinically significant and requires active treatment
12. Currently treated with a strong CYP3A4 inhibitor (e.g., erythromycin, ketoconazole, itraconazol, voriconazol, clarithromycin, telithromycin, ritonavir, mibefradil), and the treatment cannot be stopped or switched to other drug before the start of study drug administration (For a complete list, refer to this link: http://medicine.iupui.edu/flockhart/table.htm.)
13. Gastrointestinal dysfunction or gastrointestinal disease that may significantly change the absorption of study drug (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, small bowel resection, or gastric bypass)
14. History of acute pancreatitis within the past 1 year or history of chronic pancreatitis
15. Acute or chronic uncontrolled liver, pancreas or severe renal disease unrelated to the disease
16. Currently treated with a drug which may prolong QT interval, and the treatment cannot be stopped or switched to other drug before the start of study drug administration (For a complete list of products which prolong QT interval, refer to http://www.torsades.org/medical-pros/drug-lists/printable-drug-list.cfm)
17. Pregnant women, breast-feeding women

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-04; Primary Completion 2018-02 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
The rate of improvement of Dasatinib-related adverse events | at 3 months of nilotinib treatment